CLINICAL TRIAL: NCT04404959
Title: Correlation Between Perioperative Pain and Delirium in Geriatric Patients With Hip Fracture
Brief Title: Perioperative Pain and Delirium in Geriatric Patients With Hip Fracture
Acronym: Delirium-Hip
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aretaieion University Hospital (Other)
Collaborators: KAT General Hospital (Other)
Responsible Party: Principal Investigator, Dr Kassiani Theodoraki, Professor of Anesthesiology, Aretaieion University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: Delirium-Pain-Hip Fracture
Record Dates: First submitted 2020-05-22; First posted 2020-05-28 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Delirium; Delirium in Old Age; Hip Fractures; Dementia; Pain; Analgesia; Mental Status Change
MeSH Terms: conditions — Delirium; Hip Fractures; Dementia; Pain; Agnosia | interventions — Ropivacaine; Dosage Forms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fascia iliaca compartment block with ropivacaine (Active Comparator): in this arm, the fascia iliaca compartment block will be performed with 40 mL ropivacaine 0.25%
  Interventions: Other: fascia iliaca compartment block with ropivacaine
- fascia iliaca compartment block with placebo (Placebo Comparator): in this arm, the fascia iliaca compartment block will be performed with 40 mL normal saline
  Interventions: Other: fascia iliaca compartment block with placebo

INTERVENTIONS:
Other: fascia iliaca compartment block with ropivacaine — the fascia iliaca compartment block catheter will be placed with the use of ultrasound till the day of surgery. Bolus doses will be given every 12 hours (40 ml of ropivacaine 0.25%)
  Other Names: medication in regional anesthetic technique
  Arms: fascia iliaca compartment block with ropivacaine
Other: fascia iliaca compartment block with placebo — the fascia iliaca compartment block catheter will be placed with the use of ultrasound till the day of surgery. Bolus doses will be given every 12 hours (40 ml of normal saline)
  Other Names: medication in regional anesthetic technique
  Arms: fascia iliaca compartment block with placebo

SUMMARY:
The objective of this trial will be to establish whether the ultrasound-guided suprainguinal fascia iliaca compartment block is capable of protecting geriatric patients with hip fracture from delirium as compared to placebo

DETAILED DESCRIPTION:
Geriatric patients suffer from hip fractures very often. Delirium is a perioperative neuropsychiatric complication that is characterized by sudden change of mental status, inattention, disorientation and memory impairment with fluctuations of symptoms during the day. Delirium causes increased morbidity and mortality, decreased postoperative functional activity and may predispose to dementia.

Perioperative pain may be an important predisposing factor to delirium. Intravenous opioids have been widely used to relieve patients with hip fracture from pain, but they have a lot of complications and have been correlated with delirium as well. Fascia Iliaca compartment block is a peripheral compartment nerve block that is used in hip surgeries. Use of this compartment nerve block to protect geriatric patients from delirium has not been studied.

The objective of this trial will be to establish whether the ultrasound-guided suprainguinal fascia iliaca compartment block is capable of protecting geriatric patients with hip fracture from delirium as compared to placebo

ELIGIBILITY:
Inclusion Criteria:

* geriatric patients
* American Society of Anesthesiologists (ASA) I-III
* hip fracture patients

Exclusion Criteria:

* dementia
* communication or language barriers
* patients with nutritional problems
* bedridden patients

Ages: 75 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-05-10 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
pain score 30 minutes after fascia iliaca block | 30 minutes after performance of fascia iliaca block
  pain score by the use of Numeric Rating Scale (NRS) 30 minutes after fascia ilaca block, ranging from 0 to 10, where 0 means "no pain" and 10 means "worst pain imaginable"
pain score 12 hours after fascia iliaca block | 12 hours after performance of fascia iliaca block
  pain score by the use of Numeric Rating Scale (NRS) 12 hours after fascia ilaca block, ranging from 0 to 10, where 0 means "no pain" and 10 means "worst pain imaginable"

SECONDARY OUTCOMES:
pain score 1-8 days after fascia iliaca block | 1-8 days after fascia iliaca block
  pain score by the use of Numeric Rating Scale (NRS) 1-8 days after fascia ilaca block, ranging from 0 to 10, where 0 means "no pain" and 10 means "worst pain imaginable"

OTHER OUTCOMES:
Mini Mental State examination | arrival to the emergency room
  Mini Mental State examination on arrival to the emergency room
Mini Mental State examination | 1-8 days postoperatively
  Mini Mental State examination postoperatively
Confusion Assessment Method | arrival to the emergency room
  Confusion Assessment Method on arrival to the emergency room
Confusion Assessment Method | 1-8 days postoperatively
  Confusion Assessment Method postoperatively
requests for analgesia | 1-8 days postoperatively
  requests for analgesia postoperatively
tramadol consumption | 1-8 days postoperatively
  tramadol consumption postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Kassiani Theodoraki, PhD, DESA, Principal Investigator — Aretaieion University Hospital
Locations (1):
- KAT General Hospital of Athens, Kifissia, Greece

REFERENCES:
- [Background] Unneby A, Svensson PO, Gustafson PY, Lindgren APB, Bergstrom U, Olofsson PB. Complications with focus on delirium during hospital stay related to femoral nerve block compared to conventional pain management among patients with hip fracture - A randomised controlled trial. Injury. 2020 Jul;51(7):1634-1641. doi: 10.1016/j.injury.2020.04.013. Epub 2020 Apr 20. PMID 32360090
- [Background] Zhao X, Yuan W. Perioperative Multicomponent Interdisciplinary Program Reduces Delirium Incidence in Elderly Patients With Hip Fracture. J Am Psychiatr Nurses Assoc. 2022 Mar;28(2):154-163. doi: 10.1177/1078390320915250. Epub 2020 Apr 13. PMID 32281905
- [Background] Poeran J, Cozowicz C, Zubizarreta N, Weinstein SM, Deiner SG, Leipzig RM, Friedman JI, Liu J, Mazumdar M, Memtsoudis SG. Modifiable factors associated with postoperative delirium after hip fracture repair: An age-stratified retrospective cohort study. Eur J Anaesthesiol. 2020 Aug;37(8):649-658. doi: 10.1097/EJA.0000000000001197. PMID 32251149
- [Background] Uysal AI, Altiparmak B, Yasar E, Turan M, Canbek U, Yilmaz N, Gumus Demirbilek S. The effects of early femoral nerve block intervention on preoperative pain management and incidence of postoperative delirium geriatric patients undergoing trochanteric femur fracture surgery: A randomized controlled trial. Ulus Travma Acil Cerrahi Derg. 2020 Jan;26(1):109-114. doi: 10.14744/tjtes.2019.78002. PMID 31942744
- [Background] Scurrah A, Shiner CT, Stevens JA, Faux SG. Regional nerve blockade for early analgesic management of elderly patients with hip fracture - a narrative review. Anaesthesia. 2018 Jun;73(6):769-783. doi: 10.1111/anae.14178. Epub 2017 Dec 26. PMID 29278266